CLINICAL TRIAL: NCT06224244
Title: A Prospective Phase II Trial of an Accelerated Hypofractionated Radiotherapy Schedule With Risk-adapted Simultaneous Integrated Boost (HF-SIB) in Early Breast Cancer Patients Undergoing Breast Conserving Surgery
Brief Title: External Hypofractionated Radiotherapy With Simultaneous Integrated Boost in Early Breast Cancer Patients
Acronym: ESIBIRE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Silvia Takanen, Principal Investigator, Regina Elena Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1652/22
Record Dates: First submitted 2024-01-15; First posted 2024-01-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Breast Neoplasms; Breast Cancer
Keywords: Breast cancer; simultaneous integrated boost; hypofractionated radiotherapy; whole breast radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Two test groups. Phase 2 study because of 2 test groups with 2 types of SIB. A Simultaneous integrated boost to 40 Gy (SIB 40): 34 Gy to the ipsilateral breast with concomitant boost to 40 Gy to the tumor bed. A Simultaneous integrated boost to 43 Gy (SIB 43): 34 Gy to the ipsilateral breast with concomitant boost to 43 Gy to the tumor bed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simultaneous integrated boost to 40 Gy (SIB 40) (Active Comparator): Patients with the following clinico-pathological characteristics
  * pTis G3,
  * pT1 pN0/pN1mic, G1-G3 luminal biology or Her-2 positive
  Interventions: Radiation: Ten-fraction hypofractionated breast radiotherapy with 40 Gy simultaneous integrated bed boost
- Simultaneous integrated boost to 43 Gy (SIB 43) (Active Comparator): Patients with the following clinico-pathological characteristics:
  * Triple negative disease,
  * pT2 pN0/pN1mic,
  * ≤ 50 years not Luminal A
  Interventions: Radiation: Ten-fraction hypofractionated breast radiotherapy with 43 Gy simultaneous integrated bed boost

INTERVENTIONS:
Radiation: Ten-fraction hypofractionated breast radiotherapy with 40 Gy simultaneous integrated bed boost — Patients undergo BCS followed by ten-fraction adjuvant breast irradiation (34Gy) with a risk adapted SIB dose of 40 Gy
  Other Names: SIB40
  Arms: Simultaneous integrated boost to 40 Gy (SIB 40)
Radiation: Ten-fraction hypofractionated breast radiotherapy with 43 Gy simultaneous integrated bed boost — Patients undergo BCS followed by ten-fraction adjuvant breast irradiation (34Gy) with a risk adapted SIB dose of 43 Gy
  Other Names: SIB43
  Arms: Simultaneous integrated boost to 43 Gy (SIB 43)

SUMMARY:
This is a prospective non randomized phase two trial evaluating the feasibility of a ten fraction accelerated hypofractionated radiotherapy schedule with simultaneous integrated boost risk adapted in patients undergoing breast conserving surgery for early breast cancer

DETAILED DESCRIPTION:
Patients enrolled for the study, according to eligibility criteria, undergo breast conserving surgery followed by adjuvant 10-fraction whole breast irradiation with a risk adapted simultaneous-integrated boost dose at the level of the tumour bed according to clinical and pathological risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven invasive or in situ unifocal adenocarcinoma of the breast
* Breast conserving surgery
* Pathological pTis G3, pT1-2 any Grade, pN0 or pN0(sn) (isolated tumor cells [i+] allowed) pN1mic, M0 stage
* Postoperative negative (no ink) final surgical margins
* Patient requires a whole breast radiotherapy plus a tumor bed boost
* Female patients aged ≥ 18 years of any menopausal status
* ECOG performance status 0-2

Exclusion Criteria:

* Past history of malignancy except basal cell skin cancer and CIN cervix uteri or non-breast malignancy allowed if treated with curative intent and at least 5 years' disease free
* Mastectomy
* Concomitant chemotherapy (primary or sequential chemotherapy allowed) (Chemotherapy and radiotherapy must be separated by a minimum of 2 weeks). (Patients receiving neo-adjuvant chemotherapy are not excluded)
* Known disorders associated with a higher risk for complications following radiotherapy such as collagen vascular disease, dermatomyositis, systemic lupus erythematosus or scleroderma
* Any psychological, familiar, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Any serious uncontrolled medical disorder, non-malignant systemic disease, or active uncontrolled infection. Example include but are not limited to uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction or uncontrolled major seizure disorder
* Pregnant or lactating patients
* Presence of ipsilateral breast implant
* Prior breast or thoracic radiotherapy for any condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Late Effects Normal Tissue Task Force (LENT)-Subjective, Objective, Management, Analytic (SOMA) scale | From the end of treatment at 3 years
  Incidence of grade 2-3 late toxicity in terms of skin toxicity

SECONDARY OUTCOMES:
Incidence of local tumor relapse, distant metastasis and assessment of overall survival | Time from the date of the diagnosis of primary breast cancer to the date of diagnosis of local relapse, distant metastasis or death from any cause, assessed up to 60 months
  Identification of local tumor relapse in the breast parenchyma within boost volume, breast parenchyma within volume receiving 34Gy; identification of distant metastasis and analysis of overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Regina Elena Cancer Institute, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coles CE, Haviland JS, Kirby AM, Griffin CL, Sydenham MA, Titley JC, Bhattacharya I, Brunt AM, Chan HYC, Donovan EM, Eaton DJ, Emson M, Hopwood P, Jefford ML, Lightowlers SV, Sawyer EJ, Syndikus I, Tsang YM, Twyman NI, Yarnold JR, Bliss JM; IMPORT Trial Management Group. Dose-escalated simultaneous integrated boost radiotherapy in early breast cancer (IMPORT HIGH): a multicentre, phase 3, non-inferiority, open-label, randomised controlled trial. Lancet. 2023 Jun 24;401(10394):2124-2137. doi: 10.1016/S0140-6736(23)00619-0. Epub 2023 Jun 8. PMID 37302395
- [Background] Pinnaro P, Giordano C, Farneti A, Faiella A, Iaccarino G, Landoni V, Giannarelli D, Vici P, Strigari L, Sanguineti G. Short course hypofractionated whole breast irradiation after conservative surgery: a single institution phase II study. J Exp Clin Cancer Res. 2017 Dec 27;36(1):191. doi: 10.1186/s13046-017-0640-z. PMID 29282078
- [Background] Pinnaro P, Soriani A, Landoni V, Giordano C, Papale M, Marsella A, Marucci L, Arcangeli G, Strigari L. Accelerated hypofractionated radiotherapy as adjuvant regimen after conserving surgery for early breast cancer: interim report of toxicity after a minimum follow up of 3 years. J Exp Clin Cancer Res. 2010 Jan 25;29(1):9. doi: 10.1186/1756-9966-29-9. PMID 20100335